CLINICAL TRIAL: NCT03769103
Title: Open Label, Multicenter, Phase II Study of Patients With Treatment Naïve Metastatic Epidermal Growth Factor Receptor (EGFR) Mutation-Positive Non-Small Cell Lung Cancer (NSCLC) With Brain Metastases Randomized to Stereotactic Radiosurgery (SRS) and Osimertinib or Osimertinib Alone
Brief Title: Study of Osimertinib + SRS vs Osimertinib Alone for Brain Metastases in EGFR Positive Patients With NSCLC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: AstraZeneca (Industry); Princess Margaret Hospital, Canada (Other); Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LUOSICNS
Record Dates: First submitted 2018-12-03; First posted 2018-12-07 (Actual); Last update posted 2024-10-31 (Actual); Status verified 2024-10

CONDITIONS: Lung Cancer Non-small Cell Stage IV; Brain Metastases
Keywords: EGFR positive; Osimertinib; SRS
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms | interventions — osimertinib; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- SRS + Osimertinib (Active Comparator): Stereotactic radiotherapy will be delivered in 1-5 fractions to each brain metastases according to the volume and location of the metastases and clinician discretion. Osimertinib will start 1-7 days post radiotherapy.
  Interventions: Drug: Osimertinib; Radiation: Stereotactic radiotherapy
- Osimertinib alone (Experimental): Osimertinib 80mg PO daily
  Interventions: Drug: Osimertinib

INTERVENTIONS:
Drug: Osimertinib — Daily oral osimertinib
Radiation: Stereotactic radiotherapy — 1-5 fractions of stereotactic radiotherapy
  Arms: SRS + Osimertinib

SUMMARY:
This open-label, multicenter, randomized phase II study will evaluate the usage of osimertinib alone for brain metastases compared to SRS and osimertinib in patients with newly diagnosed, treatment naiive EGFR positive lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Able to provide written informed consent by patient or legally acceptable representative
* Meets the criteria in the approved regulatory indication for first line treatment with osimertinib and agree to the restrictions, monitoring, and dose-adjustment criteria stipulated in the associated product label
* Epidermal growth factor receptor (EGFR) exon 19 deletions or exon 21 (L858R) substitution mutations (either alone or in combination with other EGFR mutations)
* No prior systemic therapy except neoadjuvant, adjuvant or concurrent chemotherapy given greater than 3 months prior to enrollment on study
* Asymptomatic or minimally symptomatic brain metastases (ie. Headache, nausea, or seizure responsive to dexamethasone/analgesic/antiepileptic on stable doses of medications for a minimum of 3 days)
* Brain metastases must meet the following criteria on a diagnostic MRI: at least one lesion can be classified as measurable disease per RANO-BM, ≤ 10 brain or brainstem metastases, ≤ 30 mm and brainstem metastases must be ≤ 5 mm, metastases > 5 mm from the optic nerve or chiasm
* ECOG performance status 0-2
* Life expectancy > 6 months
* Willing to abstain from sexual activity or willing to use double-barrier method during sexual intercourse

Exclusion Criteria:

* Previous treatment with osimertinib, or any other EGFR TKI
* Patient with symptomatic brain metastases causing any neurologic deficit (not including headache, nausea, or medically controlled seizure)
* Multiple sclerosis
* Pacemaker or MRI-incompatible metal in the body
* Allergy to gadolinium MRI contrast
* Brain metastasis requiring surgery for decompression
* Leptomeningeal disease
* Previous cranial RT, or surgery for brain metastases
* Uncontrolled systemic lupus erythematosis, scleroderma or other connective tissue disorders considered a contraindication for radiotherapy
* Active cancer from another anatomical site within 5 years (non-melanomatous skin and cervical cancers permitted)
* Any medical or non-medical issue that would render patient unable to reliably complete regular QOL and neurocognitive assessments
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions and requirements
* Treatment with an investigational drug within five half-lives of the compound or 3 months, whichever is greater
* Patients with symptomatic CNS metastases who are neurologically unstable
* Patients currently receiving (or unable to stop use prior to receiving the first dose of study treatment) medications or herbal supplements known to be potent inducers of cytochrome P450 (CYP) 3A4
* Patients taking any drugs that are known to prolong QT interval that can't be withdrawn prior to Osimertinib
* Pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-03-19 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Intracranial progression free survival | 1 year
  Absence of progressive brain metastases according to the Response Assessment in Neuro-Oncology Brain Metastasis (RANO-BM criteria)

SECONDARY OUTCOMES:
Intracranial overall response rate | 2 years
  partial or complete response to therapy based on RANO-BM criteria
Time to whole brain radiotherapy (WBRT) | 2 years
  time from randomization to WBRT
Time to stereotactic radiosurgery (SRS) | 2 years
  time from randomization to SRS (not including initial SRS in the SRS + osimertinib treatment arm)
Rate of radionecrosis | 2 years
  according to institutional standards based on radiologic findings with or without pathologic confirmation and multidisciplinary review when required
Overall survival | 2 years
  defined as time from randomization to death by any cause
Time to distant progression | 2 years
  time from randomization to progression of extracranial metastases or development of new sites of disease per RECIST 1.1
Quality of life | 2 years
  Assessed by European Organisation for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) C30. Subscales for: general presence of symptoms in patients with cancer question 1-28 (1=Not at all; 4=very much); overall health/quality of life question 29-30 (1=very poor; 7=excellent) & EORTC-QLQ Brain Neoplasm (BN)20: Subscales for presence of symptoms in patients with brain tumours question 31-50 (1=Not at all; 4=very much)
Neurocognitive function | 2 years
  Assessed by Montreal Cognitive Assessment. Total score:30. 1=poor function; 30=good function
Exposure to osimertinib | 2 years
  Osimertinib dose (40mg or 80mg) for x number of days (max=730 days)

CONTACTS AND LOCATIONS:
Overall Officials: Shilo V Lefresne, MD, FRCPC, Principal Investigator — BC Cancer, Vancouver Centre; Cheryl Ho, MD, FRCPC, Principal Investigator — BC Cancer, Vancouver Centre
Locations (3):
- Canada (3):
  - BC Cancer, Vancouver Centre, Vancouver, British Columbia
  - Princess Margaret Hospital, Toronto, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Lee CK, Lefresne S, Soon YY, Robledo K, Nichol A, Sahgal A, Pinkham MB, Melosky B, Huang Y, McDermott R, Tham IWK, Parmar A, Tey JCS, Liu M, Solomon BJ, Sacher A, Leong CN, Laskin J, Koh WY, Menjak IB, Ang Y, Shultz DB, Low JL, Doherty M, Yong C, Lim MC, Tan AP, Soo RA, Hegi-Johnson F, Ho C. Osimertinib and Stereotactic Radiosurgery for Brain Metastases in EGFR-Mutated Lung Cancer: The STARLET Joint Analysis of OUTRUN and LUOSICNS Randomized Trials. J Thorac Oncol. 2026 Jan 12:103549. doi: 10.1016/j.jtho.2026.01.001. Online ahead of print. PMID 41534788